CLINICAL TRIAL: NCT04743245
Title: A Post Approval Study to Evaluate the Delivery of Hyperoxemic Super Saturated Oxygen Therapy for 60 Minutes in Anterior AMI Patients Compared to PCI
Brief Title: Delivery SSO2 Therapy for 60 Min in Anterior MI Patients With PCI ≤ 6 Hours of Symptoms Onset Compared to Standard.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TherOx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMIHOT III 09 November 2021
Record Dates: First submitted 2021-01-25; First posted 2021-02-08 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Acute Myocardial Infarction; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PCI with SSO2 therapy (Experimental): AMI subjects treated with SSO2 Therapy following PCI with stenting
  Interventions: Device: TherOx DownStream System; Device: PCI
- anterior AMI patients treated with PCI and stenting within 6 hours (Active Comparator): Control group receiving PCI with stenting alone
  Interventions: Device: PCI

INTERVENTIONS:
Device: TherOx DownStream System — SSO2 Therapy with Therox downstream System after Percutaneous Coronary Intervention (PCI)
  Arms: PCI with SSO2 therapy
Device: PCI — Standard Care of PCI

SUMMARY:
A multi-center randomized post-approval evaluation of delivery of intracoronary hyperoxemic supersaturated Oxygen therapy for 60 minutes in anterior AMI patients with successful reperfusion (via PCI) within 6 hours after onset of symptoms compared to standard therapy

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized (1:1) study. Subjects who present with anterior STEMI requiring stent placement in the proximal and/or mid LAD who meet all inclusion and exclusion criteria and provide informed consent will be treated with PCI with stenting, and if successful and uncomplicated then immediately randomized to post-procedure infusion of SSO2 Therapy for a duration of 60 minutes or standard of care.

ELIGIBILITY:
Inclusion Criteria:

-

Pre-PCI:

1. The subject must be ≥18 years of age.
2. AMI must be anterior (ST-segment elevation >1 mm in two or more contiguous leads between V1 and V4 or new left bundle branch block).
3. The subject or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided and signed written informed consent, approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC).
4. Subject and his/her physician agree to all required follow-up procedures and visits.

   ANGIOGRAPHIC INCLUSION CRITERIA: These are evaluated after the subject has provided signed Informed Consent and has undergone cardiac catheterization and PCI if indicated:
5. Based on coronary anatomy, PCI is indicated for revascularization of the culprit lesion(s) with use of a commercially available coronary stent (bare metal or drug-eluting, at operator discretion) in the LAD.
6. The primary stented infarct-related lesion(s) must be in the proximal and/or mid-LAD coronary artery (other lesions in the LAD target vessel, including diagonal branches, may be treated if clinically indicated).
7. Successful angioplasty is completed <6 hrs from symptom onset, as documented by 30% diameter residual angiographic stenosis within all treated culprit lesions with TIMI 2 or 3 flow and no major complications such as perforation or shock.
8. Expected ability to place the SSO2 delivery catheter in the coronary ostium of the left main coronary system to deliver SSO2 Therapy with stable, coaxial alignment.
9. Systemic arterial pO2 greater than or equal to 80 mmHg as measured by arterial blood gas (may be repeated if low after supplemental O2 administration).

Exclusion Criteria:

-

Patients will be excluded if ANY of the following conditions apply:

GENERAL EXCLUSION CRITERIA

Pre-PCI:

1. Prior CABG surgery.
2. Prior myocardial infarction or known prior systolic dysfunction (e.g. due to cardiomyopathy); this criterion does not include left ventricular dysfunction induced by the acute MI.
3. An elective surgical procedure is planned during the first 30 days post-enrollment.
4. Subjects who previously underwent coronary stent implantation and in whom coronary angiography demonstrates stent thrombosis to be the cause of the anterior AMI.
5. Subjects who have previously undergone an angioplasty or stenting procedure in the left anterior descending coronary artery.
6. Contraindication to MRI imaging, including any of the following:

   1. Non-MRI compatible cardiac pacemaker or implantable defibrillator;
   2. Non-MRI compatible aneurysm clip or other metallic implants;
   3. Neural Stimulator (i.e., TENS unit);
   4. Any implanted or magnetically activated device (insulin pump);
   5. Any type of non-MRI compatible ear implant;
   6. Metal shavings in the orbits;
   7. Any indwelling metallic foreign body, shrapnel, or bullet;
   8. Any condition contraindicating MRI, including claustrophobia;
   9. Inability to follow breath hold instructions or to maintain a breath hold for >15 seconds; and
   10. Known hypersensitivity or contraindication to gadolinium contrast.
7. Known impaired renal function (creatinine clearance <30 ml/min/1.73 m2 by the MDRD formula) or on dialysis.
8. Known platelet count <100,000 cells/mm3 or >700,000 cells/mm3 or a known Hgb <10 g/dL.
9. Subject has active bleeding or a history of bleeding diathesis or coagulopathy (including heparin induced thrombocytopenia), or refusal to receive blood transfusions if necessary.
10. History of intracerebral mass, aneurysm, arteriovenous malformation, or hemorrhagic stroke.
11. Stroke or transient ischemic attack within the past six (6) months, or any permanent neurological defect.
12. Gastrointestinal or genitourinary bleeding within the last two (2) months, or any major surgery (including CABG) within six weeks of enrollment.
13. Subject has received any organ transplant or is on a waiting list for any organ transplant.
14. Subject has other medical illness (e.g., cancer, dementia) or known history of substance abuse (alcohol, cocaine, heroin, etc.) that may cause non-compliance with the protocol, confound the data interpretation, or is associated with life expectancy of less than one year.
15. Subject has a known hypersensitivity or contraindication to any of the required study medications or contrast that cannot be adequately premedicated.
16. Subjects presenting with or developing in the cath lab prior to completion of the PCI procedure any of the following conditions: cardiogenic shock (SBP <80 mmHg for >30 minutes), or requiring IV pressors or emergent placement of an intra-aortic balloon pump (IABP), Impella, or other hemodynamic support for hypotension treatment, or cardiopulmonary resuscitation for >10 minutes, or ventricular fibrillation or tachycardia requiring cardioversion or defibrillation.
17. Severe known cardiac valvular stenosis or insufficiency, pericardial disease, or cardiomyopathy.
18. Subject is a member of a vulnerable population or has any significant medical or social condition which in the investigator's opinion may interfere with the subject's participation in the study or ability to comply with follow-up procedures, including MRI (e.g. alcoholism, dementia, lives far from the research center, etc.).
19. Current participation in other investigational device or drug study that has not reached its primary endpoint.
20. Previous enrollment in this study.
21. Subject is currently hospitalized for definite or suspected COVID-19.
22. Subject has previously been symptomatic with or hospitalized for COVID-19 unless he/she has been discharged (if hospitalized) and asymptomatic for ≥8 weeks and had returned to his/her prior baseline (pre-COVID) clinical condition.
23. Subject is asymptomatic (never ill) and COVID-19 PCR/antigen or antibody test is positive within the prior 4 weeks unless subject remained asymptomatic for≥4 weeks after the last positive test.

    ANGIOGRAPHIC EXCLUSION CRITERIA: These are evaluated after the subject has provided signed Informed Consent and has undergone cardiac catheterization and PCI if indicated:
24. Treatment during the index procedure of any lesion in either the left main, LCX (including the ramus), and/or RCA.
25. Post-index procedure planned intervention within 7 days (i.e., PCI of non-target lesions in any vessel, or CABG). Note: Planned revascularization (PCI or bypass) of a non-target lesion >7 days following the index procedure and after performance of the 2-7day MRI is allowed.
26. Anterior MI is due to thrombosis within or adjacent to a previously implanted stent.
27. Left ventriculography (mandatory before or after PCI, but in all cases before randomization) demonstrates severe mitral regurgitation, a ventricular septal defect, a pseudoaneurysm, aortic dissection or other mechanical complications of MI.
28. Any left main coronary artery stenosis >20%.
29. Any untreated LAD or diagonal branch lesion is present with diameter stenosis > 50% in a vessel with reference vessel diameter > 2.0 mm (visually estimated).
30. Presence of a non-stented coronary dissection with NHLBI grade >B upon completion of the PCI procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
1-year rate of Net Adverse Clinical Events (NACE) | 12 months
  The composite NACE endpoint includes a hierarchical total of the following events:
  * Death (all-cause)
  * Reinfarction
  * Target Vessel Revascularization (ischemia-driven)
  * TIMI major or minor bleeding
  * New onset heart failure or re-hospitalization for heart failure
  * Stent thrombosis (ARC definite or probable)

SECONDARY OUTCOMES:
Difference in infarct size between SSO2 Therapy and standard therapy in patients | At 2-7 days and at 6 month
  Change from 2-7 days to 6 months in MRI endpoints

CONTACTS AND LOCATIONS:
Overall Officials: James Blankenship, MD, Principal Investigator — University of New Mexico; Gregg Stone, MD, Study Chair — MOUNT SINAI HOSPITAL; Amir S Lotfi, MD, Study Director — Baystate Health
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No